CLINICAL TRIAL: NCT00920192
Title: A Phase 1/2, Open-Label, Multicenter Study of GSK1363089Gin Adult Subjects With Hepatocellular Carcinoma
Brief Title: Safety Study of Foretinib (GSK1363089) in Adults With Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111645
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: c-MET; VEGFR2; Advanced hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — GSK 1363089

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Foretinib (Experimental): Phase I starting dose of 30 mg/day escalated to 45 mg/day, de-escalated to 30 mg/day; MTD for Phase II was 30 mg/day
  Interventions: Drug: Foretinib

INTERVENTIONS:
Drug: Foretinib — Phase I starting dose 30 mg/day escalated to 45 mg/day; de-escalated to 30 mg/day. MTD for Phase II dose was 30 mg/day,

SUMMARY:
The purpose of this study is to assess the safety and tolerability of foretinib (also known as GSK1363089) when used in the treatment of patients with advanced hepatocellular carcinoma (liver cancer).

DETAILED DESCRIPTION:
The purpose of this study is to identify the maximum tolerated dose (MTD) of foretinib (also known as GSK1363089) when used in the treatment of patients with advanced hepatocellular carcinoma (liver cancer), and to assess the safety and tolerability of that dose in this patient population.

The MTD will be identified during Phase I, by standard dose-escalation of foretinib. Then Phase II will assess the safety and tolerability of foretinib dosed at MTD.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 18 years or older
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Has histologically or cytologically confirmed advanced (unresectable and/or metastatic) hepatocellular carcinoma (HCC).
* Has adequate organ system function
* Has at least 1 target tumor lesion.
* Has the ability to swallow and retain oral medication
* Has a life expectancy of at least 12 weeks
* If male:

Agrees to use double-barrier contraception, OR Agrees to complete abstinence from sexual intercourse for 14 days before exposure to investigational product, during the clinical trial, and for at least 21 days after the last dose of investigational product

- If female: Is of nonchildbearing potential OR Is of childbearing potential and has a negative serum pregnancy test within 14 days before the first dose of study drug, and agrees to use adequate contraception.

Exclusion Criteria:

* Has previously used an investigational agent or licensed drug that inhibits multiple receptor tyrosine kinases
* Is currently receiving cancer therapy
* Is currently receiving treatment with an investigational agent, including an investigational anticancer agent
* Has a Child-Pugh score >6
* Has AEs due to investigational drugs or other medications administered more than 21 days before enrollment that have not recovered to Grade 1 or less with the exception of alopecia greater than Grade 1
* Has received local therapy within the following timeframes and the subject has not fully recovered from the prior therapy: Radiotherapy: less than 28 days since completion of prior radiotherapy Chemoembolization, hepatic arterial embolization, percutaneous ethanol injection, or cryoablation: less than 42 days since completion of prior therapy Radiofrequency ablation: less than 60 days since completion of prior therapy Surgery: (1) prior surgical procedure affecting absorption, and (2) less than 28 days since last prior major surgery
* Has a history or clinical evidence of central nervous system metastases or leptomeningeal carcinomatosis
* Has a history of malabsorption syndrome, any medical condition significantly affecting gastrointestinal function, or resection of the stomach or small bowel
* Has active peptic ulcer disease, inflammatory bowel disease, or other gastrointestinal condition increasing the risk of perforation, or history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* Has a known immediate or delayed hypersensitivity or idiosyncratic reaction to drugs chemically related to foretinib.
* Has a QTcB (Bazett-corrected QT interval) or QTcF (Frederica-corrected QT interval) greater than or equal to 470 msec (or 500 msec if the subject has bundle branch block).
* Has a history of any one of the following cardiac conditions or procedures within the past 6 months: Cardiac angioplasty or stenting Myocardial infarction Unstable angina
* Has a history of a cerebrovascular accident within the past 6 months
* Has Class III or IV heart failure as defined by the New York Heart Association functional classification system
* Has poorly controlled hypertension (systolic blood pressure of 140 mm Hg or greater or diastolic blood pressure of 90 mm Hg or greater)
* Has a history of untreated deep venous thrombosis within the past 6 months (e.g., calf vein thrombosis)
* Has a history of main portal vein thrombosis
* Has the presence of any nonhealing wound, fracture, or ulcer, or the presence of symptomatic peripheral vascular disease
* Has had previous or concurrent cancer that is distinct in primary site or histology from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (tumor stages Ta, Tis, and T1). Any cancer curatively treated more than 3 years before study entry is permitted.
* Has a history of bleeding varices within the past 30 days
* Has had clinically significant gastrointestinal bleeding within the past 30 days
* Is a pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08-12 (Actual); Primary Completion 2012-03-07 (Actual); Study Completion 2015-03-24 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) | up to 2 years
Safety and tolerability of foretinib at the MTD as measured by number and severity of AEs | up to 2 years

SECONDARY OUTCOMES:
The antitumor activity of foretinib at the MTD according to RECIST | up to 2 years
PK profile of foretinib | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- GSK Investigational Site, Hong Kong, Hong Kong
- Taiwan (2):
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Singh RP, Patel B, Kallender H, Ottesen LH, Adams LM, Cox DS. Population pharmacokinetics modeling and analysis of foretinib in adult patients with advanced solid tumors. J Clin Pharmacol. 2015 Oct;55(10):1184-92. doi: 10.1002/jcph.546. Epub 2015 Jul 7. PMID 25998042
- See also: Results for study 111645 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111645?search=study&search_terms=111645#rs
- Available data/document: Statistical Analysis Plan: 111645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111645 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register